CLINICAL TRIAL: NCT06615297
Title: Demonstration of the Relationship Between Mimic Muscle Volume and Central Facial Palsy Severity and Dysphagia
Brief Title: Mimic Muscle Volume, Central Facial Palsy Severity and Dysphagia
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-40
Record Dates: First submitted 2024-09-13; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Facial Paralysis, Central; Stroke
MeSH Terms: conditions — Facial Paralysis; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- central facial paralysis: 70 stroke patients with central facial paralysis who were included in the rehabilitation program at Istanbul Physical Therapy and Rehabilitation Training and Research Hospital will be included
  Interventions: Diagnostic Test: ultrasonographic evaluation

INTERVENTIONS:
Diagnostic Test: ultrasonographic evaluation — facial nerve thickness (right/left), depressor labi inferior, depressor anguli oris, buccinator and risorius muscles will be evaluated.

SUMMARY:
70 stroke patients with central facial paralysis will be included and their demographic data will be questioned and facial nerve thickness, depressor labi inferior, depressor anguli oris, buccinator and risorius muscles will be evaluated.

DETAILED DESCRIPTION:
70 stroke patients with central facial paralysis who were included in the rehabilitation program at Istanbul Physical Therapy and Rehabilitation Training and Research Hospital will be included and their demographic data such as age, gender, marital status, education level, body mass index, stroke etiologies will be questioned and used with the House-Brackmann scale. Involvement levels, facial nerve thickness (right/left), depressor labi inferior, depressor anguli oris, buccinator and risorius muscles will be evaluated. The data obtained will be correlated with total dysphagia score and facial disability index.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke and presence of unilateral central facial paralysis,
* Agreeing to participate in the study,
* Cognitive competence to understand the test instructions,
* Presence of communication skills to respond to the test instructions.

Exclusion Criteria:

* Presence of previous facial paralysis or a neurological disease other than stroke that will cause central paralysis,
* bilateral involvement
* illiteracy, refusal to participate in the study,
* jaw joint problem,
* surgical intervention in the facial area that will affect ultrasound measurements,
* infected open wound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 stroke patients with central facial paralysis who were included in the rehabilitation program at Istanbul Physical Therapy and Rehabilitation Training and Research Hospital will be included
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
facial nerve thickness | baseline
  the thickness of the nerve will be measured by ultrasound

SECONDARY OUTCOMES:
depressor labi inferior | baseline
  the thickness of the muscle will be measured by ultrasound
depressor anguli oris | baseline
  the thickness of the muscle will be measured by ultrasound

IPD SHARING:
Plan to Share IPD: Undecided